CLINICAL TRIAL: NCT01202539
Title: Use of Real-time Infrared Reflective Marker Tracking and Surface Texture Mapping to Assess the Integrity of a Novel Thermoplastic Mask System for Frameless Immobilization
Brief Title: Real-time Assessment of Frameless Intrafraction Motion
Status: Withdrawn | Type: Observational
Why Stopped: Enrollment challenges
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, James A. Tanyi, Principal Investigator, Oregon Health and Science University
Other Study IDs: OHSU IRB00006460
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to assess the ability of a modified thermoplastic mask system in keeping an individual head stationary for a predefined amount of time. The investigators hope to know if the modified mask is study enough, and also if the modification on the mask will allow the investigator see and track the individual's movement underneath the mask by means of a camera that can detect light reflected from the individual. Participants will lay down on their backs and their heads will be held in place with the mask system for approximately 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individual
* Age > 18 years.
* Males and females of all races and ethnic groups

Exclusion Criteria:

* Severe claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential subjects will be recruited by the Oregon Health and Science University study investigators.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: James A. Tanyi, Ph.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- See also: Oregon Health and Science University — http://www.ohsu.edu